CLINICAL TRIAL: NCT02333851
Title: Comparison of Basal-bolus and Premixed Insulin Regimens in Hospitalized Patients With Type 2 Diabetes (PININ Study)
Brief Title: Basal-bolus and Premixed Insulin Regimens in Hospitalized Patients With Type 2 Diabetes (PININ Study)
Acronym: PININ
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Safety reasons
Sponsor: Hospital Universitario Central de Asturias (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDOHUCA1
Record Dates: First submitted 2014-12-20; First posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus treatment; Hospitalized patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin, pork; isophane insulin, pork drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Premixed insulin (Experimental): Mixtard 30:70 Novonordisk® twice daily, before breakfast and before dinner.
  Interventions: Drug: Mixtard 30:70 Novonordisk® twice daily
- Basal-bolus (Experimental): 'Lantus® once daily and Apidra® before meals
  Interventions: Drug: Lantus® once daily and Apidra® before meals

INTERVENTIONS:
Drug: Mixtard 30:70 Novonordisk® twice daily — Premixed insulin twice daily before breakfast and before dinner
  Other Names: Premixed 30:70 insulin two times a day
  Arms: Premixed insulin
Drug: Lantus® once daily and Apidra® before meals — Injection of Lantus® insulin once daily and rapid insulin Apidra® before breakfast, lunch and dinner
  Other Names: Basal bolus regimen
  Arms: Basal-bolus

SUMMARY:
Pilot study to compare the efficacy and safety of a premixed-insulin regimen (70% intermediate insulin and 30% regular insulin) to a basal-bolus insulin regimen (glargine once daily and glulisine before meals) hospitalized patients with type 2 diabetes.

DETAILED DESCRIPTION:
Pilot, randomized, prospective, open-label study admitted to the Hospital with a previous diagnosis of type 2 diabetes or with a blood glucose level on admission greater than 180 mg/dl.

Patients were randomized to receive a premixed human insulin formulation with 70% intermediate insulin plus 30% regular insulin (Mixtard 30®, Novo Nordisk) or a basal-bolus regimen with glargine once daily and glulisine before meals (Lantus® and Apidra®, Sanofi-Aventis).

The primary outcome of the study was to determine differences in glycemic control between treatment groups as measured by mean daily blood glucose concentration during the hospital stay. Secondary objectives were to determine differences in the percentage of glucose measures between 80 and 180 mg/dl, frequency and severity of hypoglycemic events, total daily insulin use, length of hospital stay and glycemic viability between groups.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of type 2 diabetes with a blood glucose level on admission greater than 180 mg/dl and treated with diet, any combination of oral antidiabetics agents and/or insulin therapy

Exclusion Criteria:

* Patients with hyperglycemia without a previous diagnosis of diabetes
* Patients with acute hyperglycemic emergencies or with severe hyperglycemia treated with intravenous insulin infusion on admission
* Patients with acute or chronic kidney disease (serum creatinine greater than 2 mg/dl),
* Patients treated with corticosteroids
* Patients with history of severe or repeated hypoglycemic episodes
* Pregnant women
* Patients expected to require ICU admission or less than 3 days of hospital stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Differences in mean daily blood glucose concentration | Participants will be followe for the duration of hospital stay, an expected average of 2 weeks
  Glucose concentration were measured in capillary blood 6 times a day, before and 2 hours after meals and daily mean calculated

SECONDARY OUTCOMES:
Number and severity of hypoglycemia episodes | Participants will be followe for the duration of hospital stay, an expected average of 2 weeks
  Frequency and severity of hypoglycemia episodes during all the stay in the hospital
Measures of dispersion of glycemia values (Glycemia variability) | Participants will be followe for the duration of hospital stay, an expected average of 2 weeks
  Glycemia variability will be measured by standard deviation of blood glucose values, coefficient of variation and mean amplitude of glycemic excursions or MAGE.
Total daily Insulin use in International Units per Kg of weight | Participants will be followe for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edelmiro Menéndez Torre, Principal Investigator — Hospital Universitario Central de Asturias